CLINICAL TRIAL: NCT00615563
Title: Utilization of HIV Drug Resistance Testing in Treatment Experienced Patients (UTILIZE Study)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Other Study IDs: 1182.116
Record Dates: First submitted 2008-01-31; First posted 2008-02-14 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- genotype test
  Interventions: Behavioral: NO BI Drug administered
- combined phenotype/genotype test
  Interventions: Behavioral: NO BI Drug administered

INTERVENTIONS:
Behavioral: NO BI Drug administered

SUMMARY:
The primary objective of this trial was to assess the presence of susceptibility to tipranavir and other ARVs of the HIV-1 isolates in treatment experienced patients. The secondary objective was to examine clinicians' use of HIV drug resistance testing in treatment experienced patients currently failing a PI based HAART regimen.

ELIGIBILITY:
Inclusion criteria

Patients that meet the following inclusion criteria will be eligible for participation in this study:

1. Signed patient informed consent prior to study participation.
2. HIV-1 infected male or female ?18 years of age.
3. Have confirmed (2 consecutive) HIV RNA ?1000 copies/mL (one of the results must be within 3 months of enrollment into the study).
4. Current HAART regimen contains a protease inhibitor for ?3 months.
5. Physicians considering a change in the patient?s HAART regimen. f.) History of treatment with 2 or more protease inhibitors (including the current PI). Low dose ritonavir (i.e.< 400 mg. bid) is not counted as one of the PIs.

Exclusion criteria

A patient with any of the following criteria will be excluded from participation in the study:

1. ARV medication naive.
2. Active opportunistic infection. c.) Known or suspected non-adherence to current HAART regimen as assessed by the investigator.

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01

PRIMARY OUTCOMES:
Level of sensitivity of a patient's HIV-1 isolate to tipranavir | Day 1
Levels of sensitivity of a patient's HIV-1 isolate to other marketed ARVs (PIs, NRTIs, and NNRTIs). | Day 1

SECONDARY OUTCOMES:
Protease inhibitor(s) (PI) identified by the clinician prior to resistance testing to which a patient's HIV-1 virus was thought to be susceptible | Day 1
PI that was discontinued or initiated after receiving resistance testing results | up to 45 days
Non-PI ARVs that were discontinued or initiated after receiving resistance testing results | up to 45 days
Rationale reported for modifying or not modifying baseline ARV regimen after receiving resistance testing results | up to 45 days
Utilization (yes/no) of expert interpretation by a clinician after receiving resistance testing results | up to 45 days
Relationship between prior number of PIs utilized and number of available (sensitive) PIs as determined by resistance testing | up to 45 days
The physician's assessment of whether the phenotypic testing (as part of combined testing) provided more information than the genotypic test alone did | up to 45 days
Physician reported limitations that influence access to resistance testing | day 1
Clinician reported reasons why tipranavir was or was not considered as an option for each patient | up to 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharmaceuticals,Inc./Ridgefield
Locations (31):
- United States (30):
  - Boehringer Ingelheim Investigational Site, Bakersfield, California
  - Boehringer Ingelheim Investigational Site, Beverly Hills, California
  - Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - Boehringer Ingelheim Investigational Site, Los Angeles, California
  - Boehringer Ingelheim Investigational Site, Newport Beach, California
  - Boehringer Ingelheim Investigational Site, Oakland, California
  - Boehringer Ingelheim Investigational Site, Stanford, California
  - Boehringer Ingelheim Investigational Site, Daytona Beach, Florida
  - Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - Boehringer Ingelheim Investigational Site, Miami, Florida
  - Boehringer Ingelheim Investigational Site, North Palm Beach, Florida
  - Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - Boehringer Ingelheim Investigational Site, Berkley, Michigan
  - Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - Boehringer Ingelheim Investigational Site, Camden, New Jersey
  - Boehringer Ingelheim Investigational Site, Newark, New Jersey
  - Boehringer Ingelheim Investigational Site, Voorhees Township, New Jersey
  - Boehringer Ingelheim Investigational Site, Rochester, New York
  - Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - Boehringer Ingelheim Investigational Site, Huntersville, North Carolina
  - Boehringer Ingelheim Investigational Site, Akron, Ohio
  - Boehringer Ingelheim Investigational Site, Portland, Oregon
  - Boehringer Ingelheim Investigational Site, Dallas, Texas
  - Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - Boehringer Ingelheim Investigational Site, Houston, Texas
  - Boehringer Ingelheim Investigational Site, Hampton, Virginia
- Boehringer Ingelheim Investigational Site, Ponce, Puerto Rico